CLINICAL TRIAL: NCT00179751
Title: A Phase I/II Study Of Lenalidomide (Revlimid ) In Combination With Gemcitabine In Patients With Untreated Advanced Carcinoma Of The Pancreas
Brief Title: A Phase I/II Study of Lenalidomide in Combination With Gemcitabine in Patients With Untreated Advanced Carcinoma of the Pancreas
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Collaborators: Prologue Research International (Industry)
Organization: Celgene (Industry)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-PANC-001
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2005-11-07 (Estimated); Status verified 2005-11

CONDITIONS: Pancreatic Cancer
Keywords: cc-5013; revlimid; pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Lenalidomide; Gemcitabine

INTERVENTIONS:
Drug: CC-5013
Drug: gemcitabine

SUMMARY:
Phase I will determine the MDT and evaluate the safety profile of oral lenalidomide days 1-21 and weekly gemcitabine days 1, 8, & 15 in 28 day cycles Phase II will explore the anti-tumor activity and safety of the combination in subjects with advanced pancreatic carcinoma. Subjects will receive oral lenalidomide days 1-21 and weekly gemcitabine days 1, 8, & 15 in 28 day cycles until documented disease progression occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must understand and voluntarily sign an informed consent document.
2. Age >or = to 18 years at the time of signing informed consent form.
3. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
4. Histological documentation of advanced pancreatic carcinoma not amenable to curative surgery or definitive radiation.
5. Radiographic or clinical evidence of measurable advanced pancreatic carcinoma. Subjects must have measurable disease at least 2 cm in diameter.
6. Subjects may have been previously treated with radiation therapy and 5-fluorouracil as a radiosensitizer in the adjuvant setting if they currently have evidence of progression.
7. ECOG performance status of 0 or 1 (Appendix I: ECOG Performance Status Scale).
8. Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 7 days of starting study drug. In addition, sexually active WCBP must agree to use adequate contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on study medication.

Exclusion Criteria:

1. Any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) <1,500 cells/mm3 (1.5 x 109/L)
   2. Platelet count <100,000 cells/mm3 (100 x 109/L)
   3. Serum creatinine >2.5 mg/dL (221 mmol/L)
   4. Serum SGOT/AST or SGPT/ALT >3.0 x upper limit of normal (ULN)
   5. Serum total bilirubin >2.0 mg/dL (34 mmol/L)
2. Any serious medical condition or psychiatric illness that places the subject at an unacceptable risk for study participation or would prevent the subject from signing the informed consent.
3. Prior history of malignancy (except basal cell or squamous cell carcinoma or carcinoma in situ of the breast) unless the subject has been free of disease for > or = to 1 year.
4. Known brain or leptomeningeal disease (CT scan or MRI of the brain required only in case of clinical suspicion of central nervous system involvement).
5. Prior use of systemic therapy for the treatment of carcinoma of the pancreas with the exception of 5-fluorouracil as a radiosensitizer in the adjuvant setting.
6. Concurrent use of any other anti-cancer agents.
7. Any prior use of lenalidomide.
8. Prior > or = to grade 3 (see Appendix III) allergic reaction/hypersensitivity to thalidomide.
9. Prior > or = to grade 3 (see Appendix III) rash or any desquamating (blistering) rash while taking thalidomide.
10. Use of any standard/experimental anti-cancer drug therapy within 28 days of the initiation of study drug therapy.
11. Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-04; Study Completion 2006-08

PRIMARY OUTCOMES:
Phase I-To determine the maximum tolerated dose (MTD) and evaluate the safety profile of oral lenalidomide days 1- 21 in combination with gemcitabine days 1, 8, and 15 every 28 days in subjects with advanced pancreatic carcinoma.
Phase II-To explore the anti-tumor activity of the combination of lenalidomide on days 1 - 21 and gemcitabine days 1, 8, and 15 every 28 days in subjects with advanced pancreatic carcinoma.

SECONDARY OUTCOMES:
Phase I-To explore the anti-tumor activity of the combination of lenalidomide and gemcitabine as combination therapy in subjects with advanced pancreatic carcinoma.
Phase II-To evaluate the safety profile of the combination of lenalidomide and gemcitabine as combination therapy in subjects with advanced pancreatic carcinoma.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cancer and Blood Institute, Metairie, Louisiana
  - Bernard Cancer Center, St Louis, Missouri
  - Case Western Reserve University Hospitals Ireland Cancer Center, Cleveland, Ohio
  - Charleston Cancer Center, Charleston, South Carolina
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas